CLINICAL TRIAL: NCT06642519
Title: Adaptive Cortical Neuromodulation Using a Brain-machine Interface to Treat Freezing of Gait in Parkinson's Disease.
Brief Title: Brain-Machine Interface for Freezing of Gait
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Alfonso Fasano, Professor, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-5435
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease; Freezing of Gait Symptoms in Parkinson's Disease
Keywords: Brain-Machine interface; Freezing of Gait; Triggered stimulation; Adaptive Stimulation
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ECoG implantation (Experimental): Patients will be implanted with high-density cortical ECoG arrays during DBS surgery.
  Interventions: Other: Brain Stimulation

INTERVENTIONS:
Other: Brain Stimulation — Studies will be conducted using ECoG, with a bidirectional interface, both recording (aim/phase 1) and stimulating (aim/phase 2), during real-world gait and FOG in PD patients over the course of 7-days of gait experiments.

SUMMARY:
Gait problems in Parkinson's disease (PD), especially freezing of gait (FOG), greatly affect quality of life. While deep brain stimulation (DBS) is a highly effective treatment for many motor symptoms of PD, it is less effective for, or can even worsen, gait issues. The primary motor cortex (M1) plays a crucial role in the network that controls gait, particularly in initiating movement. Changes in local field potentials (LFPs) from the subthalamic nucleus (STN) are associated with different aspects of gait. However, detecting abnormal brain activity related to FOG requires a method called electrocorticography (ECoG), which has revealed that during FOG, there is increased beta-gamma phase amplitude coupling (PAC) in the M1.

Brain-machine interfaces (BMIs) have shown promise in understanding motor functions by decoding brain activity. It is believed that BMIs could provide both accurate indicators of FOG and targeted treatments for it in PD.

Our objectives are to use a high-density ECoG-based BMI to both record and stimulate brain activity during real-world gait and FOG in PD patients who are undergoing standard DBS procedures. Our goals are to improve our understanding of the brain's role in FOG and normal gait in PD and to develop new treatments based on cortical stimulation.

Aim 1 - Identify gait biomarkers: brain activity from the M1/SMA cortex during different phases of walking and during FOG episodes, both with and without medication will be recorded. Machine learning will be used to identify the brain patterns linked to FOG.

Aim 2 - Use cortical stimulation to stop FOG: Cortical stimulation and its effects on leg and trunk movements will be studied by measuring muscle activity, movement, and posture during different states, such as resting, standing, walking, and during FOG episodes. The type of stimulation which is most effective at stopping FOG will be identified.

ELIGIBILITY:
Inclusion Criteria:

* PD fulfilling standard criteria for bilateral STN/GPi DBS surgery
* Debilitating FOG in the off-medication condition with only partial response to levodopa (defined as the witnessed occurrence of FOG during the on phase of the pre-DBS L-dopa challenge)
* Clinically established FOG (i.e. reported by patient/caregiver AND seen by the examiner in the clinic)
* Able to provide informed consent, comply with study protocol

Exclusion Criteria:

* Prior ischemic stroke, intracranial hemorrhage, or intracerebral mass
* Previous brain surgery
* Other disorders potentially biasing assessment
* Absence of FOG in the medication on condition (a population already manageable with current standard of treatment).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Number and Duration FOG episodes | 7-day experiment
  The number and duration of FOG episodes either with or without stimulation, including the number/duration of FOG episodes with optimal stimulation.

SECONDARY OUTCOMES:
Measurement of Chronic Coupling between Cortex and Basal Ganglia | 7-day experiment
  The aim is to explore the chronic coupling between cortex and basal ganglia by means of deep brain recordings. This is an exploratory opportunity that will be pursued while carrying out the main aims. However, DBS electrodes will not be turned on to provide stimulation until after they exit the study, after which regular standard-of-care DBS programming will occur.
Exploring BMI Control to Trigger and Study FOG | 7-day experiment
  It has never been established if individuals with FOG display typical or impaired performance in brain-machine interfaces (BMI) control and whether they can experience phenomena similar to FOG while performing these virtual tasks. This is also an exploratory aim. Participants will be trained to guide virtual effectors (cursors) on a screen using the implanted BMI. The aim is to stablish if standard BMI tasks can trigger FOG-like phenomena. Such occurrence would largely augment the possibility of testing new neuromodulation paradigms to prevent and abolish FOG in laboratory settings.

CONTACTS AND LOCATIONS:
Locations (1):
- Movement Disorders Centre - Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided